CLINICAL TRIAL: NCT05712291
Title: Optimization of Total Knee Arthroplasty Using Robotic Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 199617
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-09

CONDITIONS: Knee Osteoarthritis
Keywords: total knee arthroplasty; robotic total knee arthroplasty; the active robotic surgical system; robotic system in orthopedic
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total knee arthroplasty using the active robotic system (Other): Total knee arthroplasty using the active robotic surgical system TSolution One TCAT, and system for planning TPlan
  Interventions: Procedure: Total knee arthroplasty using the active robotic surgical system; Device: TSolution One TCAT, and system for planning TPlan
- total knee arthroplasty using the standard manual technic (Other): Primary total knee arthroplasty using the standard recommended set of instruments
  Interventions: Procedure: total knee arthroplasty using the standard manual technic

INTERVENTIONS:
Procedure: Total knee arthroplasty using the active robotic surgical system — Total knee arthroplasty using the active robotic surgical system TSolution One TCAT, and system for planning TPlan
  Arms: total knee arthroplasty using the active robotic system
Device: TSolution One TCAT, and system for planning TPlan — the active robotic surgical system TSolution One TCAT, and system for planning TPlan
  Arms: total knee arthroplasty using the active robotic system
Procedure: total knee arthroplasty using the standard manual technic — total knee arthroplasty using the standard manual technic
  Arms: total knee arthroplasty using the standard manual technic

SUMMARY:
For the first time, it is planned to create algorithms for working with a robotic system at different patient flow rates, optimize the use of computed tomography to assess bone density and pronounced osteophytes, develop an algorithm and tactics for treating bilateral osteoarthrosis of the knee joint using an active robotic system. Aim: optimization of total knee arthroplasty using robotic systems and improvement of treatment outcomes. Objectives: to develop algorithms for preoperative planning, surgical intervention using an active robotic system; to improve the technique of active robotic total knee arthroplasty in osteoporosis, osteosclerosis and pronounced osteophytes; to develop a tactic for the treatment of patients with bilateral osteoarthrosis of the knee joint using an active robotic system. It is planned to conduct an open-label retrospective and prospective clinical study in parallel observations.The study is planned to include 250 patients with osteoarthritis of the knee joint stage 3-4 (according to Kellgren-Lawrence). The methodology developed and improved in the dissertation will be introduced into the work of the clinical Departments of Traumatology, Orthopedics and Disaster Surgery, studying the learning curve.

DETAILED DESCRIPTION:
Relevance: Robotic orthopedic surgery has been around for over twenty years and is becoming more relevant every day. Modern systems consist of a robotic arm, robotic cutting tools and robotic milling systems with a variety of navigation systems with using active, semi-automatic or passive control systems. In the analysis of clinical studies, it can be concluded that these robotic systems reduce variability and increase the accuracy of positioning and alignment of prosthesis components. A new generation of robotic systems is currently being actively introduced into the field of arthroplasty interventions, which can eliminate pain and improve the quality of life of patients with end-stage osteoarthritis of the knee joint.

Total knee arthroplasty (TKA) in the terminal stages of gonarthrosis is one of the most effective and technologically advanced operations. More than 700,000 surgeries are performed annually in the United States and the number continues to grow. According to the literature in Russia for 2011-2019. out of 27,906 TKAs, the proportion of primary arthroplasties was 92.3% (n = 25,759). It should be noted that the number of operations of primary knee arthroplasty increased almost 2 times - from 1678 in 2011 up to 3,730 in 2019. Therefore, TKA is attracting attention from many manufacturers of robotic surgical systems.

With the introduction of an active robotic system into clinical practice, a number of problems have arisen: high time costs of perioperative actions; the operation of an active robotic unit with high or low bone density, pronounced osteophytes; operation of an active robotic unit in bilateral TKA.

The novelty of the proposed topic: For the first time in Russia it is planned to create algorithms for working with a robotic system at different patient flow rates, optimize the use of computed tomography to assess bone density and pronounced osteophytes, develop an algorithm and tactics for treating bilateral osteoarthrosis of the knee joint using an active robotic system.

Aim and objectives of the research:

Aim: optimization of total knee arthroplasty using robotic systems and improvement of treatment outcomes.

Objectives: to develop algorithms for preoperative planning, surgical intervention using an active robotic system; to improve the technique of active robotic total knee arthroplasty in osteoporosis, osteosclerosis and pronounced osteophytes; to develop a tactic for the treatment of patients with bilateral osteoarthrosis of the knee joint using an active robotic system.

Type of new research: an open-label, retrospective and prospective observational clinical study in parallel groups.

Research object and number of observations: the study is planned to include 250 patients with osteoarthritis of the knee joint of stage 3-4 (according to Kellgren-Lawrence).

Methods of the research:

1. General clinical examination of patients (collection of complaints, examination, assessment of physical findings and local status);
2. Assessment of the range of motion in the knee joint before and after surgery;
3. Performing X-ray images and CT of the knee joint before and after surgery, with the determination of the angles: HKA, LDFA, MPTA, Q; Preoperative 3D planning on the TPLAN workstation; Surgical treatment. 1) Primary total knee arthroplasty using the active robotic surgical system TSolution One, TCAT.

Evaluation of patient treatment results according to scales: VAS, KSS, OKS, WOMAC, ASA, FJS-12.

Methods of statistical processing of the material: statistical processing of data is planned to be carried out on a personal computer using Excel software packages and using standard methods of variation statistics using SPSS 16 statistical software packages.

Estimated research result:

Algorithms of actions for preoperative planning and surgical intervention will be developed.

An approach will be developed for the diagnosis, classification and treatment of patients with pronounced areas of osteosclerosis of the knee joint during robotic total knee arthroplasty.

An approach will be developed for the diagnosis and treatment of patients with concomitant osteoporosis in robotic total knee arthroplasty.

A tactic for the treatment of patients with bilateral osteoarthritis of the knee joint of stage 3-4 (according to Kellgren-Lawrence) will be proposed.

The methodology developed and improved in the dissertation will be introduced into the work of the clinical bases of the Department of Traumatology, Orthopedics and Disaster Surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of written informed consent of the patient to participate in the study;
2. Patients with stage 3-4 osteoarthritis of the knee joint (according to Kellgren-Lawrence).
3. Men and women from 21 to 90 years old.
4. Pain in the knee joint above 3 points according to VAS
5. Opportunity for observations during the entire study period (12 months);
6. Mental adequacy, ability, willingness to cooperate and to fulfill the doctor's recommendations.

Exclusion Criteria:

1. Refusal of the patient from surgical treatment;
2. Presence of contraindications to surgical treatment;
3. Severe forms of diabetes mellitus (glycosylated hemoglobin> 9%);
4. Diseases of the blood (thrombopenia, thrombocytopenia, anemia with Hb <90 g / l);
5. The patient's unwillingness to conscious cooperation.
6. Refusal of the patient to participate in the study;
7. Non-compliance with the hospital regimen, according to the order of the Ministry of Health and Social Development of Russia dated 01.08.07, No. 514;
8. The impossibility of observing the patient within the control period after the operation.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Implant position assessment | 2 months after surgery
  CT scanning; these diagnostic methods assess the position of the implant, analysis of deformation, assessment of the angles in the knee joint (LDFA, MPTA, MA, these diagnostic methods assess the position of the implant, analysis of deformation, assessment of the angles in the knee joint, analyze the rotation of implant)
Implant position assessment | 6 months after surgery
  CT scanning
Implant position assessment | 12 months after surgery
  CT scanning

SECONDARY OUTCOMES:
Quality of life and knee function assessment | 2,6,12 months after surgery
  Knee Society Score(KSS score), which combines subjective and objective information and separates the knee score (pain, stability, range of motion etc.) from the functional score of the patient (ability to walk, go up and down stairs)
Quality of life assessment (joint awareness after surgery) | 2,6,12 months after surgery
  FJS-12, measures the clinical outcomes focusing on joint awareness after surgery
Quality of life assessment (the condition of patients) | 2,6,12 months after surgery
  WOMAC score is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints
Pain assessment | 2,6,12 months after surgery
  Visual Analog Score (VAS) for pain - dynamics pain assessment
Quality of life assessment (an individual's activities of daily living) | 2,6,12 months after surgery
  OKS score. The OKS is a patient reported outcome measure that consists of 12 questions about an individual's activities of daily living and how they have been affected by pain over the preceding four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Gritsyuk, PhD, Study Chair — The First MSMU (I.M.Sechenov).The Department of Traumatology, Orthopedics
Locations (1):
- University clinical hospital №1 I.M.Sechenov First Moscow State Medical University. The Department of Traumatology, Orthopedics and Disaster Surgery, Moscow, Russia

REFERENCES:
- [Background] LYCHAGIN A.V.1, a, GRITSYUK A.A.1, b, RUKIN Y.A.1, c, ELIZAROV M.P.1, d, THE HISTORY OF THE DEVELOPMENT OF ROBOTICS IN SURGERY AND ORTHOPEDICS (LITERATURE REVIEW). 2020; 1 (39)2020: 10.17238/issn2226-2016.2020.1.13-19
- [Background] LYCHAGIN A.V. 1, a, RUKIN Y.A. 1, b, GRITSYUK A.A. 1, c, ELIZAROV M.P. 1, d, FIRST EXPERIENCE OF USING AN ACTIVE ROBOTIC SURGICAL SYSTEM IN TOTAL KNEE ARTHROPLASTY. 2019; 4 (38) 2019: 10.17238/issn2226-2016.2019.4.27-33